CLINICAL TRIAL: NCT03458065
Title: Myocardial Injuries and Hemodynamic Stress Biomarkers: a Comparison Between Transvenous and Subcutaneous ICD Shock
Brief Title: T-ICD vs S-ICD Shocks: Myocardial Injuries
Acronym: MYSTIC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Monaldi Hospital (Other)
Responsible Party: Principal Investigator, Antonio D'Onofrio, MD, FESC, Monaldi Hospital
Other Study IDs: MonaldiH
Record Dates: First submitted 2018-03-01; First posted 2018-03-08 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: ICD Shock Myocardial Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- S-ICD
  Interventions: Device: ICD
- T-ICD
  Interventions: Device: ICD

INTERVENTIONS:
Device: ICD — Implantable Cardioverter Defibrillator

SUMMARY:
Implantable cardioverter defibrillator (ICD) shocks are associated with a subsequent increased risk of death, and an elevation of cardiac enzymes has been measured after defibrillation testing (DFT). The aim of our study was to investigate the association between S-ICD vs T-ICD shocks and acute cardiac damage in humans, as evaluated by means of sensitive and highly specific circulating biomarkers

ELIGIBILITY:
Inclusion Criteria:

patients who met the criteria for ICD implantation according to the current guidelines

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who met the criteria for ICD implantation according to the current guidelines
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2018-09-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
myocardial micro-damage | 6 months
  degree of myocardial micro-damage, assessed by calculating the variation in the serum levels of high-sensitivity cardiac troponin I (hs-CTnI) and creatine kinase-MB mass concentration (CK-MB mass), measured before and after an S-ICD shock delivered during intraoperative DFT

CONTACTS AND LOCATIONS:
Locations (1):
- Monaldi Hospital, Naples, Italy

IPD SHARING:
Plan to Share IPD: No